CLINICAL TRIAL: NCT06773611
Title: Electronic Register on Advanced Heart Failure and Transplantation
Brief Title: Electronic Register on Advanced Heart Failure and Transplantation di Cuore
Status: Recruiting | Type: Observational
Sponsor: IRCCS Azienda Ospedaliero-Universitaria di Bologna (Other)
Responsible Party: Sponsor
Other Study IDs: Rescat
Record Dates: First submitted 2025-01-09; First posted 2025-01-14 (Actual); Last update posted 2025-01-14 (Actual); Status verified 2024-12

CONDITIONS: Heart Failure; Heart Transplantation
MeSH Terms: conditions — Heart Failure

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Patient Registry: Yes
Target Follow-Up Duration: 5 Years
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The goal of this observational study is to create an electronic registry of patients diagnosed with Advanced Heart Failure or Heart Transplant, starting from 01/01/1985 and to assess the incidence of Advanced Heart Failure and Heart Transplant, and characterize patients affected by the first or undergoing the second procedure, starting from 01/01/1985. The primary outcomes are:

* Hospitalization for cardiovascular cause
* Death

DETAILED DESCRIPTION:
Heart failure is a pathological condition characterized by high morbidity and mortality, and it leads to a significant worsening of the quality of life for patients. The treatment of heart failure involves various options; the goal is to slow down the progression of the disease, reduce hospitalizations, increase survival, and reduce symptoms in order to improve the quality of life. Treatments range from pharmacological therapy to lifestyle changes, from device implantation to heart transplant surgery. Early diagnosis and treatment often help reduce symptoms, and many patients with heart failure can return to an active life. Patients with heart failure must undergo regular check-ups to assess their general physical condition and the status of the disease. It is therefore essential to evaluate and systematize the different therapies.

This study is both retrospective and prospective

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years
* Ability to provide informed consent
* Diagnosis of Advanced Heart Failure or Heart Transplant

Exclusion Criteria:

* none

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All adult patients attending the SSD Heart Failure and Transplants unit of the IRCCS Azienda Ospedaliero-Universitaria di Bologna will be evaluated, starting from 01/01/1985. Each patient has been and will be followed according to standard care practices.
Sampling Method: Non-Probability Sample
Enrollment: 10000 (Estimated)
Dates: Start 2023-09-04 (Actual); Primary Completion 2028-09 (Estimated); Study Completion 2028-09 (Estimated)

PRIMARY OUTCOMES:
Hospitalization for cardiovascular cause | 5 years
  Hospitalization for cardiovascular cause
Death | 5 years
  Death

SECONDARY OUTCOMES:
Hospitalization for non-cardiovascular cause | 5 years
  Hospitalization for non-cardiovascular cause
Implantation of medical device (including mechanical support) | 5 years
  Implantation of medical device (including mechanical support)
Need for intravenous diuretic therapy | 5 years
  Need for intravenous diuretic therapy
Need for hemodialysis event | 5 years
  Need for hemodialysis event

CONTACTS AND LOCATIONS:
Overall Officials: Luciano G Potena, MD, Principal Investigator — IRCCS Azienda Ospedaliero-Universitaria di Bologna
Locations (1):
- IRCCS Azienda Ospedaliero-Universitaria di Bologna, Bologna, Italy